CLINICAL TRIAL: NCT01467375
Title: An Open Label, Non Comparative, Multicentre Extension Trial to Assess the Long Term Safety and Efficacy of Biphasic Insulin Aspart 30 in Subjects With Type 2 Diabetes Who Have Completed BIAsp-1234
Brief Title: Long Term Safety and Efficacy of Biphasic Insulin Aspart 30 in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-1361
Record Dates: First submitted 2011-11-04; First posted 2011-11-08 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: biphasic insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart — Individually adjusted dose, injected s.c. (under the skin) before breakfast and dinner

SUMMARY:
This trial is conducted in Oceania and North America. The aim of this trial is to assess the long term safety and efficacy of biphasic insulin aspart 30 in subjects with type 2 diabetes who have completed the BIAsp-1234 trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have been correctly included in and completed BIAsp-1234

Exclusion Criteria:

* Persistent non-compliance with study medication, visit schedules or other trial specific procedures during the preceding trial
* Fulfilment of any withdrawal criteria prior to and including the final visit of the BIAsp-1234.
* Females only: breast feeding, intention of becoming pregnant, or judged to be using inadequate contraceptive measures (adequate contraceptive methods are sterilisation,IUD (Intra Uterine Device), oral contraceptives or barrier methods)
* Known or suspected allergy to trial product or related products
* Development since entry into the previous trial of late diabetic micro or macro vascular complications, which in the opinion of the Investigator indicates a progressed state of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2001-01-08 (Actual); Primary Completion 2004-10-22 (Actual); Study Completion 2004-10-22 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events
Frequency of hypoglycaemic episodes

SECONDARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (12):
- Australia (8):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Parkville, Victoria
  - Novo Nordisk Investigational Site, Ashford
  - Novo Nordisk Investigational Site, Auchenflower
  - Novo Nordisk Investigational Site, Launceston
  - Novo Nordisk Investigational Site, Nowra
  - Novo Nordisk Investigational Site, Ringwood
  - Novo Nordisk Investigational Site, Rooty Hill
- Canada (4):
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Québec
  - Novo Nordisk Investigational Site, Saskatoon

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com